CLINICAL TRIAL: NCT05118698
Title: An Intervention Study of Gynostemma Pentaphyllum in Patients With Metabolic Syndrome
Brief Title: Explore the Effect of Gynostemma Pentaphyllum on Patients With Metabolic Syndrome
Acronym: GPMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJTU1AF2021LSK-273
Record Dates: First submitted 2021-10-15; First posted 2021-11-12 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose group (Experimental): Participants will be allowed to drink Gynostemma pentaphyllum powder containing 12% saponin, 2 g each time, 3 times a day for 3 months.
  Interventions: Drug: Gynostemma
- Low-dose group (Experimental): Participants will be allowed to drink Gynostemma pentaphyllum powder containing 8% saponin, 2 g each time, 3 times a day for 3 months.
  Interventions: Drug: Gynostemma
- Placebo group (Placebo Comparator): Participants will be allowed to drink a placebo of spinach powder with almost no saponin content, 2 g each time, 3 times a day for 3 months.
  Interventions: Other: Spinach

INTERVENTIONS:
Drug: Gynostemma — Patients in the high-dose group and low-dose group will take gynostemma powder with a saponin content of 12% and 8% respectively, 3 times a day for 3 months.
  Arms: High-dose group; Low-dose group
Other: Spinach — For the spinach powder group, each patient will take spinach powder with nearly no saponin content, 3 times a day for 3 months.
  Arms: Placebo group

SUMMARY:
Previous research shows that gypenoside could keep blood lipid and blood sugar under control in an effective way. In this study, we intend to explore whether gypenosides have clinical improvement effects on metabolic diseases such as diabetes, hyperlipidemia, and non-alcoholic fatty liver and their cardiovascular protective potential. It is designed to recruit 150 patients with metabolic syndrome diagnosed who meet the criteria for enrollment, and randomly divide them into three groups. Gynostemma powder, with two different saponins content (12% and 8%) from Pingli County, Shaanxi Province, and spinach powder with almost no saponins were used to conduct the intervention on patients. Patients will be followed up regularly at the beginning of each month from the first enrollment until the third month. At each follow-up, data of patient's anthropometric indicators as well as clinical inspection indicators related to metabolism (blood routine, liver function, etc.) will be recorded. In addition, patient's blood, hair, urine, and stool samples will be collected to further explore the mechanism of diseases.

ELIGIBILITY:
Inclusion Criteria:

* Low-density lipoprotein (LDL) cholesterol ≥130 mg/dL (3.4 mmol/L ), or conforms to the diagnosis criteria for metabolic syndrome (based on the MetS diagnostic criteria developed by IDF and AHA in 2009), that is, having three or more of the following traits:

  1. waist circumference ≥90 cm in men or ≥80 cm in women;
  2. Elevated TG (drug treatment for elevated TG is an alternate indicator) ≥150 mg/dL (1.7 mmol/L);
  3. Reduced HDL-c (drug treatment for reduced HDL-c is an alternate indicator) < 40 mg/dL (1.03 mmol/L) in males < 50 mg/dL (1.29 mmol/L) in females;
  4. Elevated blood pressure (anti-hypertensive drug treatment in a patient with a history of hypertension is an alternate indicator). Systolic ≥ 130 and/or diastolic ≥ 85 mmHg;
  5. Elevated fasting glucose (drug treatment for elevated glucose is an alternate indicator) ≥ 100 mg/dL (5.6 mmol/L).
* Be over 18 years old or younger than 80 years old, no gender limit.
* Have a good follow-up compliance and can be followed up for more than 3 months;
* From 2 weeks before enrollment to the end of the entire trial, the treatment regimen will not change.

Exclusion Criteria:

* Pregnant and lactating women;
* Allergic or toxic reactions to gynostemma and other drugs;
* Infectious diseases such as viral hepatitis, AIDS, syphilis, tuberculosis are active;
* After drug treatment, still showing high blood sugar (fasting blood glucose higher than 200mg/dL, 11.1mmol/L) or hyperlipidemia, or hypertension (higher than 180/110 mmHg);
* Any conditions judged by the investigator that affect enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
change of weight | From date of randomization to the last follow-up, once a month, assessed up to 3 months.
  Kg
change of blood lipid level | From date of randomization to the last follow-up, once a month, assessed up to 3 months.
  mmol/L
change of blood glucose level | From date of randomization to the last follow-up, once a month, assessed up to 3 months.
  mmol/L

SECONDARY OUTCOMES:
change of waistline and hipline | From date of randomization to the last follow-up, once a month, assessed up to 3 months.
  cm
change of blood pressure | From date of randomization to the last follow-up, once a month, assessed up to 3 months.
  mmHg
change of glucose tolerance | The date of first enrollment and 3 months after the intervention.
  mmol/L
change of serum insulin level | The date of first enrollment and 3 months after the intervention.
  pmol/L
change of serum C peptide level | The date of first enrollment and 3 months after the intervention.
  pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Bingyin Shi, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China